CLINICAL TRIAL: NCT02085512
Title: Prevention of PTSD by Neurocognitive Training of Emotional Regulation
Brief Title: Prevention of PTSD III: Neurocognitive Training of Emotional Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Stanford University (Other); Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-00879
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Post Traumatic Stress Disorder; Major Depression; Anxiety Disorders
Keywords: Post Traumatic Stress Disorder (PTSD); Major Depression; Secondary Prevention; Neurocognitive Retraining; Randomized Controlled Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurocognitive retraining (Experimental): Neurobehavioral training will be delivered through the web, with prompting for training tasks accomplished through daily emails that include a single integrated log-in system using a customized implementation with OneLogin. All training tasks have "game-like" features making them visually engaging, and motivating. The training tasks provide immediate feedback about performance, and are specifically designed to target circuitry critical for executive functioning (EF) and emotional reactivity.
  Interventions: Procedure: Neurocognitive retraining Web Based Intervention
- Control, Web Based Tasks (Placebo Comparator): Engaging daily, for 30 days in web-based video games or reading tasks that do not specifically engage or train neurocognitive functions.
  Interventions: Other: Control, web-based tasks

INTERVENTIONS:
Procedure: Neurocognitive retraining Web Based Intervention — Neurobehavioral training will be delivered through the web, with prompting for training tasks accomplished through daily emails that include a single integrated log-in system using a customized implementation with OneLogin. All training tasks have "game-like" features making them visually engaging, and motivating. The training tasks provide immediate feedback about performance, and are specifically designed to target circuitry critical for executive functioning (EF) and emotional reactivity.
  Arms: Neurocognitive retraining
Other: Control, web-based tasks — No training modules
  Arms: Control, Web Based Tasks

SUMMARY:
The proposed work will evaluate the ability of neurocognitive retraining of executive functions and emotional regulation to reduce neurocognitive dysfunctions that follow trauma exposure and thereby prevent PTSD. The scientific rationale for this work is the hypothesis that impaired emotional regulation interferes with the expected recovery from the early responses to traumatic events, leading into a chronic disorder. In an initial phase the investigators will recruit 20 recently traumatized participants among trauma survivors admitted to a general hospital emergency room and test the planned intervention's acceptance and right 'dosing'. In the second phase the investigators will enroll 80 recent survivors into a randomized controlled study of the new intervention. The intervention will consist of web-based neurobehavioral training interventions that instill an emotional bias toward positive stimuli, improve emotion recognition and labeling, reduce resistance to emotional distraction, and enhance executive functioning. Control participants will complete web-based video games that do not have emotion-regulatory benefits. Outcome measures will include improvement in neurocognitive functioning and in PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult survivors of traumatic events consecutively admitted to a general hospital Emergency Department

Exclusion Criteria:

* Chronic PTSD at the time of the traumatic event. Current and lifetime psychotic or bipolar illness, current substance abuse save alcohol, medical condition precluding participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Amelioration of neurocognitive impairments that are associated with post-traumatic stress disorder | Three and nine months after a traumatic event
  Impairments in emotional reactivity, emotion regulation, and executive functioning critically contribute to post-trauma psychopathology (including, but not restricted to PTSD). The primary outcome measure of this work are changes (improvements) of these functions at the immediate aftermath of treatment and six months later

SECONDARY OUTCOMES:
Post-traumatic Stress Disorder (PTSD) symptoms | Three and nine months after a traumatic event
  Decrease in PTSD symptoms from trial's onset

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Y Shalev, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Fonzo GA, Fine NB, Wright RN, Achituv M, Zaiko YV, Merin O, Shalev AY, Etkin A. Internet-delivered computerized cognitive & affective remediation training for the treatment of acute and chronic posttraumatic stress disorder: Two randomized clinical trials. J Psychiatr Res. 2019 Aug;115:82-89. doi: 10.1016/j.jpsychires.2019.05.007. Epub 2019 May 8. PMID 31125916

DOCUMENTS (1):
  • Study Protocol (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT02085512/Prot_000.pdf